CLINICAL TRIAL: NCT05971628
Title: Resection And Partial LIver Transplantation With Delayed Hepatectomy for Hepatocellular Carcinoma
Acronym: RAPID-HCC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP210351
Record Dates: First submitted 2023-06-30; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver transplantation; split; auxiliary transplantation; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liver transplantation with the RAPID procedure (Experimental): Liver transplantation for hepatocellular carcinoma according to the RAPID protocol. This protocol is an auxiliary liver transplantation of a partial graft with total hepatectomy in two stages (2 successive operations).
  Interventions: Procedure: RAPID procedure
- Comparator group with standard liver transplantation (whole graft) (No Intervention): Orthotopic liver transplantation with whole organ from deceased donor for hepatocellular carcinoma. Data will be provided by Biomedicine Agency, following pairing rules.

INTERVENTIONS:
Procedure: RAPID procedure — RAPID procedure stands for Resection And Partial Liver Transplantation with Delayed Hepatectomy for hepatocellular carcinoma
  Arms: Liver transplantation with the RAPID procedure

SUMMARY:
This is a national, non-randomized, multicentric trial evaluating the feasibility and the tolerance of the RAPID procedure in patients with HCC with preserved liver function requiring a liver transplantation.

DETAILED DESCRIPTION:
In France, the liver transplant allocation is based on the severity of liver failure, but patients with hepatocellular carcinoma (HCC) usually do not have hepatocellular failure, resulting in reduced access to liver transplantation. Two years after registration on the LT list, only 66% of those registered are transplanted due to tumor progression. This observation leads to the paradoxical conclusion that better access to transplantation is an absolute priority, but remains limited by the shortage of grafts.

The split surgical of one graft into two grafts is the most effective way to increase the number of transplantable organs. This technique is performed daily as part of pediatric TH where the child receives the left lobe/liver, adapted to his morphology. However, in adults, transplantation of the left lobe (segments 2+3) or of the left liver (segments 2+3+4) associated with complete excision of the native liver generates a high rate of complications (small-for-size syndrome) and compromises graft and recipient survival. For these reasons, this type of procedure has been almost abandoned in France.

One of the ways to increase the organ pool without risking liver failure is therefore to perform an auxiliary transplant with a partial graft from an organ harvested in its entirety and then shared.

The investigators therefore wish to evaluate the feasibility and tolerance, the results and the "gain" of grafts after a standardized RAPID procedure ( Resection And Partial LIver Transplantation with Delayed Hepatectomy) allowing to transplant an adult with a left lobe (very small graft) from a shared whole graft (deceased donor in brain death) , and to compare the results with standard management (orthotopic HT with whole organ for HCC).

The population is 50 major patients (in order to realize the RAPID procedure for 34 patients) with HCC requiring LT according to the usual transplantability criteria, with preserved liver function. The study lasts a maximum of 70 months (24 months of inclusion period, 6 months between selection and inclusion, <12 months between inclusion and the 1st RAPID time, 4 months maximum between the 2 RAPID Steps, 24 months of patient follow-up post 2nd step of RAPID). The study will proceed as described below :

* Pre-selection, information and consent of the patient by the local team.
* After validation by the scientific committee of the inclusion/exclusion criteria, the patient will be prioritized with the Biomedicine Agency (800 points at 6 months)
* If necessary, he will receive a waiting treatment for the CHC
* Step 1 of RAPID : During the first operation, he will have a left hepatectomy and then LT with a left lobe/liver in an orthotopic position. During this operation, a treatment (resection/destruction) of a possible HCC of the right liver can be proposed in order to not to leave active nodule(s).
* Step 2 of RAPID : Within a maximum of 4 months, after graft hypertrophy, right hepatectomy of the remaining native liver will be realized.
* The oncological and post-LT follow-up will then be no different from a standard out-of-protocol patient. Standard immunosuppression
* At the end of the study, a comparative analysis will be made with the control group, the anonymous data of which will be transmitted by the ABM.

The expected benefits for participants are :

* Rapid access to LT thanks to prioritization by the Biomedicine Agency at 6 months. Moreover, prioritization on the list could make it possible to limit the use of waiting treatments (surgery, radiation therapy, chemoembolization, immunotherapy, etc.) with non-negligible side effects/morbidity (e.g. arterial dissection jeopardizing the future graft) and high costs.
* reduction in the risk of leaving the list, of death on the list,
* access to an excellent quality graft (strict donor selection criteria) while patients with HCC frequently receive marginal organs, known as "out of turn", in an attempt to reduce their wait,
* possible improvement in intention-to-treat survival.

The expected benefits for society are :

* Overall increase in the organ pool = partial response to the shortage of organs from which all recipients will be able to benefit (reduction of waiting time),
* reduction of costs related to waiting treatments in CHCs (patients registered on the list),
* reduction of costs related to hospitalization in the event of acute decompensation of chronic liver disease (ACLF).

The risks added by research :

* The main risk is that caused by two successive interventions, close together. The international literature on orthotopic auxiliary grafting using a small graft shows that the morbidity is real but the medium and long-term results are good (4 postoperative deaths reported only).
* The risk of small for size syndrome is not ruled out in the RAPID protocol but will be limited to a minimum by appropriate portal modulation measures, a surgical technique refined and implemented by the experience of each center + literature, and finally postoperative follow-up close.

ELIGIBILITY:
Inclusion criteria (RAPID receiver)

* 18 years ≤ age ≤ 68 years
* Indication of LT for HCC validated in multidisciplinary meeting
* AFP score ≤ 2 (15)
* Body mass index < 30 kg/m2
* MELD score ≤ 15, without access to prioritization
* PET CT-choline and PET CT-FDG without sign of extra-hepatic localizaton
* Patient having been informed and able to give written consent to participate in the RAPID-HCC study
* Validation of the patient's inclusion in the RAPID-HCC protocol by the scientific committee

Exclusion criteria

* History of, liver transplant, surgical or radiological portocaval anastomosis
* History of major abdominal surgery (including hepatectomy)
* History of abdominal radiotherapy (extrahepatic)
* History of acute/chronic pancreatitis
* Expected combined transplant
* HCC located 1 cm away from the transection line required by the first stage hepatectomy
* Portal or arterial thrombosis
* patient with a pre-graft hepatic venous pressure gradient ≥ 20mmHg
* Ascites (clinical or radiological) less than 5 years ago
* Hepatitis C viral load +
* Acute or chronic hepatitis B (not cured)
* HIV + serology
* Severe comorbidities, in particular severe cardiovascular or respiratory or renal pathology (at the discretion of the medical-surgical team)
* Patient on anticoagulant treatment
* Patient who has received (or is due to receive) preoperative treatment with radioembolization on the right side, hepatectomy or radiotherapy near the hilum
* Patient who received (or should receive) preoperative treatment with anti-tyrosine kinase (TKI) less than three months ago
* Patients receiving or having received immunotherapy

Donor selection criteria:

* Brain-dead donor (no living donor)
* 18 years ≤ age ≤ 65 years
* Hepatic, vascular and biliary anatomy compatible with performing a split. Analysis entrusted to the team that will carry out the split, and based on the scanner of the donor (to be available on the Biomedicine Agency website)
* Biological and hepatic assessment compatible with the realization of a split, in particular transaminases < 4 times the normal
* Graft not assigned to a protocol requiring machine infusion.
* Serology: anti-HBc negative, anti-HCV negative

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient with successful RAPID procedure | 4 months after the second RAPID step
  Success of the procedure will be assessed as a patient :
  * who complete the 2 steps of the procedure,
  * who had no graft resection and who is still alive 4 months later.
Tolerance of the RAPID procedure | from first stage of the surgical protocol and until 90 days after the second stage
  Tolerance will be assessed with Adverse events related to the procedure

SECONDARY OUTCOMES:
Proportion of grafts in place | 4 months after the first surgical step
  Number of patients with a graft in place at 4 months after the first surgical step
Survival of grafts at 2 years from liver transplantation (LT) | at 2 Years from LT
  Survival RAPID grafts considered in the event of a graft still in place Non-survival in the event of the patient's death or new LT
Survival of patient at 2 year after their registration on the waiting list of transplantation | at 2 year after their registration on the waiting list of transplantation
  whatever the cause of death
Survival of patient at 2 year after LT | at 2 year after LT
Incidence of rejection after RAPID | at 2 years after the first stage of RAPID
  Identification of histologically proven rejections within 2 years after the first stage of RAPID.
Waiting time between listing on the waiting list and LT according to RAPID | 1 year
  Time between registration the waiting list and TH according to RAPID (1st step)
Gain of grafts | 70 months
  Number of left lobes transplanted according to RAPID protocol - the number of retransplantations = organ gain obtained. Will be also analysed, the number of right livers generated and transplanted, as well as the number of complete RAPID procedures (native liver excision) will also be analyzed.
Comparison of the drop-out rate between RAPID group and control group | 18 months
  Drop out will be estimated by exclusion from the LT program, whatever the cause : death, worsening, transplant refusal, etc.
Comparison of the waiting time between registration on the transplantation list and LT between RAPID group and control group | up to 18 months
  Patients who completed the 1st RAPID phase compared to the control group
Comparison of the graft survival at 2 years after LT between RAPID group and control group | at 2 years after 1rst stage of RAPID

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GOLSE, Doctor, Principal Investigator — APHP, Paul Brousse Hospital, villejuif, France
Locations (1):
- AP-HP, Paul Brousse Hospital, Villejuif, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peloso A, Pietrasz D, Daillier E, Cylly L, Scatton O, Goumard C, Mabrut JY, Mohkam K, Lesurtel M, Dokmak S, Jeddou H, Boudjema K, Allard MA, Adam R, Sa Cunha A, Azoulay D, Cherqui D, Vibert E, Golse N. Resection and partial liver transplantation from deceased donors with delayed total hepatectomy (RAPID procedure) for hepatocellular carcinoma: a national, multicenter, non-randomized, prospective trial. BMC Cancer. 2025 May 9;25(1):848. doi: 10.1186/s12885-025-14127-7. PMID 40346479